CLINICAL TRIAL: NCT07361133
Title: Cyclophosphamide and Etoposide as a Promising Metronomic Therapy in Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Cyclophosphamide and Etoposide as a Metronomic Therapy in Advanced Head and Neck Squamous Cell Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO 2504-505-120-198
Record Dates: First submitted 2025-12-04; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma; Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Keywords: Cyclophosphamide; Etoposide; Head and neck squamous cell carcinoma; Advanced recurrent; Metastatic
MeSH Terms: conditions — Recurrence; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — Cyclophosphamide; Etoposide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide and Etoposide in combination (Experimental): Participants in intervention arm will receive cyclophosphamide IV 400 mg/m2 every 3 weeks and etoposide 100 mg/m2 daily for 3 days every 4 weeks, for total 6 months.
  Interventions: Drug: Cyclophosphamide and Etoposide in combination
- Methotrexate (Active Comparator): Participants in control arm will receive weekly Methotrexate 50 mg for total 6 months.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Cyclophosphamide and Etoposide in combination — Cyclophosphamide IV 400 mg/m2 every 3 weeks and etoposide 100 mg/m2 daily for 3 days every 4 weeks for 6 months.
  Arms: Cyclophosphamide and Etoposide in combination
Drug: Methotrexate — 50 mg weekly for 6 months
  Arms: Methotrexate

SUMMARY:
The goal of this clinical trial is to learn if drugs as cyclophosphamide (C) and etoposide (E) work to treat advanced head and neck cancer in adults. It will also learn about the safety of both drugs. The main questions it aims to answer are:

Do drugs C and E work to treat advanced head and neck cancer, after failure on first line chemotherapy? What medical problems do participants have when taking drugs C and E? Researchers will compare drugs C and E in combination to a placebo (a look-alike substance that contains no drug) to see if these 2 drugs works to treat advanced head and neck cancer.

Participants will:

Take drug C every 3 weeks and drug E every 4 weeks or a placebo every week for 6 months.

Visit the clinic once every 3 weeks for checkups and tests. Keep a diary of their symptoms.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the potential efficacy of cyclophosphamide and etoposide as metronomic therapy in recurrent/resistant and/or metastatic head and neck squamous cell carcinoma adults after failure on first line chemotherapy, or intolerant to further aggressive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, age = or > 18 years
* Participants with recurrent head and neck squamous cell carcinoma after failure on first line chemotherapy.
* Participants with advanced progressed, resistant, metastatic head and neck squamous cell carcinoma.

Exclusion Criteria:

* Adjuvant and Neoadjuvant head and neck squamous cell carcinoma patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Cyclophosphamide and Etoposide as metronomic therapy | From first day of the study to the end of treatment at 6 months.
  The efficacy of Cyclophosphamide and Etoposide as metronomic therapy in improving disease response. Tumor size (tumor dimensions: length, width, height) as measured by Computed Tomography, illustrating whether the disease is progressed, regressed or stationary. In addition to serum LDH level. Both will be assessed every 3 cycles.

SECONDARY OUTCOMES:
Assessment of clinical symptoms | From the first day of the study till the end of treatment at 6 months
  Clinical symptoms will be assessed each cycle of treatment through assessment of pain by Numeric Pain Rating Scale, difficulty in swallowing, persistent hoarseness, weight loss.
Progression free survival | From first day of the study till the end of study at 6 months
  Evaluation of the progression free survival at the end of study
Overall survival | From the first day of study till the end of study at 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participants data can not be shared for patient confidentiality.

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/j.annonc.2024.10.456